CLINICAL TRIAL: NCT02649270
Title: Single and Multiple Dose -Based Tolerability, Safety and Pharmacokinetic Phase 1 Study of Humanized Anti-CD6 Monoclonal Antibody Injection in Chinese Patients With Psoriasis
Brief Title: Tolerability, Safety and Pharmacokinetic Study of Humanized Anti-CD6 Monoclonal Antibody Injection in Chinese Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: company strategy
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-T1h-PSO-1
Record Dates: First submitted 2015-05-12; First posted 2016-01-07 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Psoriasis
Keywords: Tolerability; Safety; Pharmacokinetic Study; preliminary pharmacodynamic study; Humanized Anti-CD6 Monoclonal Antibody(T1h)
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group1 (Experimental): 10 Psoriasis patients,T1h 0.2mg/kg,only single dose administration at week 1.
  Interventions: Biological: T1h
- Group2 (Experimental): 10 Psoriasis patients,T1h 0.4mg/kg ,first administration at week 1 and continous administration from fifth week for 9 weeks.
  Interventions: Biological: T1h
- Group3 (Experimental): 10 Psoriasis patients,T1h 0.8mg/kg,first administration at week 1 and continous administration from fifth week for 9 weeks.
  Interventions: Biological: T1h
- Group4 (Experimental): 10 Psoriasis patients,T1h 1.6mg/kg,first administration at week 1 and biweekly from fifth week for 9 weeks.
  .
  Interventions: Biological: T1h

INTERVENTIONS:
Biological: T1h — Given T1h for different groups by vein to evaluate safety and tolerability;Collecting blood samples for pharmacokinetics and pharmacodynamics after administration.
  Other Names: Anti-CD6 Monoclonal Antibody

SUMMARY:
The humanized recombinant anti-CD6 monoclonal antibody Injection (T1h) has been approved for psoriasis in India. The first trial in China is to evaluate the tolerability, safety, pharmacodynamic, pharmacokinetics and preliminary efficacy of T1h for patients with psoriasis.

DETAILED DESCRIPTION:
The humanized recombinant anti-CD6 monoclonal antibody (T1h) is developed whose ligand binding properties of the original murine monoclonal antibody are preserved on the CD6 molecule. T1h monoclonal antibody has been approved for clinical studies of autoimmune diseases in Cuba and India, such as psoriasis and rheumatoid arthritis (RA).

Single and multiple dose based tolerability, safety and pharmacokinetic phase 1 Study of Humanized Anti-CD6 Monoclonal Antibody Injection in Chinese patients with psoriasis, 40 patients are enrolled. They are divided into 4 groups (0.2mg/kg, 0.4mg/kg, 0.8mg/kg, 1.6mg/kg) and each group includes 10 patients. First, these doses are all single-dose administration gradually from low then the doses 0.4mg/kg, 0.8mg/kg and 1.6mg/kg are multi-dose administration gradually from low.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 55 years, males or females ( no less than 3 patients in each dose group)
2. Patients with chronic plaque psoriasis for at least 6 months (until patients with an informed consent) with or without arthritis psoriasis
3. BSA≥3% or PASI≥10
4. PGA≥3
5. Patients were eligible if wash-out period was no less than the time as follows:

   * 2 weeks for topical retinoic acid or glucocorticoid therapy
   * 6 months for retinoic acid of this kind drugs therapy
   * 2 weeks for light therapy
   * 4 weeks for Psoralen combined with UV-A therapy
   * 4 weeks for methotrexate(MTX),cyclophosphamide,cyclosporine and other immunosuppressive therapy
   * 7 half life time periods for other systemic immunosuppressive therapy
   * 8 weeks for Biological agents for psoriasis therapy
6. Fertile males or females who are willing to adopt contraceptive methods (e.g. hormonal pitch, intrauterine device, condoms)
7. Patients were voluntary to sign a written informed consent.

Exclusion Criteria:

1. The females were pregnant, or lactating or showed positive urine pregnancy reaction during screening.
2. Patients with erythroderma or pustular psoriasis.
3. Patients receiving glucocorticoid systemic drug therapy.
4. Patients previously or currently suffered from autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome ), or suffering from primary or secondary immunodeficiency or human immunodeficiency virus
5. Patients with any active infection (nail bed induced fungal infections were excluded), chronic infections, and tuberculosis history.
6. Patients with severe heart disease, heart failure, asthma, chronic obstructive pulmonary disease or neuropsychiatric diseases.
7. Patients previously or currently suffered from tumors including solid tumors, hematologic malignancies and carcinoma in situ.
8. Patients with positive tests for hepatitis B surface antigen (HBsAg), hepatitis C serology (HCV-Ab) or human immunodeficiency virus (HIV-Ab)
9. Patients with Hemoglobin < 90 g/L, white blood cell count <3.5 × 10^9 / L, neutrophil count <1.5 × 10^9 / L, or platelet count <80 × 10^9 / L
10. Patients with more than doubled serum cereal third transaminase(ALT )and glutamic-oxaloacetic transaminase(AST) as the upper limit of the reference value or serum creatinine values were above the upper limit of the reference.
11. Patients with a history of drug abuse or alcoholism
12. Patients were allergic to a recombinant biologic agent or any component of proteins derived from murine
13. Patients with surgery within three months or any planned surgery or laser skin treatment within six months
14. Patients received any vaccination within 28 days
15. Patients received any experimental drug treatment within three months
16. Patients were not suitable determined by researchers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Adverse events | from patients with informed consents to 30 days after the last administration

SECONDARY OUTCOMES:
single-dose ,Peak plasma concentration (Cmax) of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose, Area under the plasma concentration versus time curve( AUC(0-t)) of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose, Area under the plasma concentration versus time curve(AUC(0-∞))of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose, Time to peak(Tmax) of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose,Elimination rate constant （kel）of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose,Half time (t1/2) of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose,Total body clearance (CLs)of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose,Apparent volume of distribution(Vd) of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
single-dose,Mean residence time(MRT) of T1h | -2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after administration
multiple dose,Time to peak(Tmax) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose,Peak plasma concentration in steady state(Css_max) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose,Minimum plasma concentration in steady state(Css_min) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose,Average plasma concentration in steady state(Css_avg) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose, Area under the plasma concentration versus time curve in steady state(AUCss) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose,Apparent volume of distribution in steady state (Vss) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose,Degree of fluctuation (DF) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
multiple dose,Accumulation Index(AI) of T1h | -2h,0h at week5,6,7,8,9,10,11,12;2h、-1h、-0.5h、0h、1h、2h、6h、12h、24h、2d、3d、7d、14d、21d、28d after week13
Erythrocyte sedimentation rate(ESR) | week7,9 at -2h;week13 at -2h,24h,7d,14d,21d,28d after administration
C-reactive protein(CRP) | week7,9 at -2h;week13 at -2h,24h,7d,14d,21d,28d after administration
Tumor Necrosis Factor -alpha(TNF-α) | week7,9 at -2h;week13 at -2h,24h,7d,14d,21d,28d after administration
Interleukin (il)-6 (IL-6) | week7,9 at -2h;week13 at -2h,24h,7d,14d,21d,28d after administration
interferon--γ (IFN-γ) | week7,9 at -2h;week13 at -2h,24h,7d,14d,21d,28d after administration
CD6 | week7,9 at -2h;week13 at -2h,24h,7d,14d,21d,28d after administration
Psoriasis Area and Severity Index(PASI) | at the end of 4th week,8th week,12th week after administration
Physician's Global Assessment(PGA) | The 29th day,The 57th day,The 85th day and The 113th day after administration
Body surface area(BSA) | The 29th day,The 57th day,The 85th day and The 113th day after administration

CONTACTS AND LOCATIONS:
Overall Officials: lihong liu, Principal Investigator — Beijing Chao Yang Hospital; yanling he, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China